CLINICAL TRIAL: NCT01636180
Title: Effect of the Repeated Loading Dose of Clopidogrel and High Dose of Clopidogrel Continuous Therapy on the Platelet Aggregation Inhibition in Patients With Myocardial Infarction Undergoing Interventional Treatment.
Acronym: REL-0609
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Fundacja Ośrodek Badań Medycznych (Other)
Collaborators: KCRI (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1.0, 2009-06-06
Record Dates: First submitted 2012-04-05; First posted 2012-07-10 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Acute Myocardial Infarction
Keywords: STEMI; NSTEMI; clopidogrel; Areplex; REL-0609
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction | interventions — Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clopidogrel - Repeated Loading Dose (Experimental): repeated loading dose of clopidogrel (600 mg) in addition to high dose of clopidogrel continuous therapy for 30 days (150 mg/day)
  Interventions: Drug: Clopidogrel
- Clopidogrel - standard of care (Active Comparator): no repeated loading dose of clopidogrel with clopidogrel continuous therapy for 30 days (75 mg/day)
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel — repeated loading dose of clopidogrel (600 mg) in addition to high dose of clopidogrel continuous therapy for 30 days (150 mg/day)
  Arms: Clopidogrel - Repeated Loading Dose
Drug: Clopidogrel — no repeated loading dose of clopidogrel with clopidogrel continuous therapy for 30 days (75 mg/day)
  Arms: Clopidogrel - standard of care

SUMMARY:
REL-0609 trial's hypothesis is that repeated loading doses of clopidogrel (600 mg) administration in addition to high dose of clopidogrel continuous therapy (150 mg/day) results in higher inhibition of the platelets' aggregation in patients with myocardial infarction undergoing interventional treatment comparing to the standard therapy. Such treatment strategy will not cause increased risk of bleeding complications. In many trials treatment with to repeated loading doses of clopidogrel together with high dose of clopidogrel continuous therapy resulted in: MACE reduction, improvement of the long term therapy results, lower risk of ischemic complications. Currently, data regarding to the results of the above treatment are still limited.

DETAILED DESCRIPTION:
The objectives of the study is:

* to evaluate the effect of the repeated loading dose of clopidogrel (600 mg) in addition to high dose of clopidogrel continuous therapy (150 mg/day) on the platelet aggregation inhibition in patients with myocardial infarction undergoing interventional treatment
* to evaluate the safety of the repeated loading dose of clopidogrel (600 mg) in addition to high dose of clopidogrel continuous therapy (150 mg/day) in patients with myocardial infarction undergoing interventional treatment

ELIGIBILITY:
Inclusion Criteria:

•≥18 years of age,

* Myocardial Infarction with or without ST segment elevation,
* clopidogrel treatment (confirmed administration of loading dose of 600 mg or chronic therapy of 75 mg/day),
* signed written informed consent.

Exclusion Criteria:

* prior administration of fibrinolytic therapy and/or GP IIb/IIIa inhibitors within the last 14 days,
* prior administration of prasugrel within the last 14 days,
* subject with known hypersensitivity to the active ingredient or other components of the product
* increased risk of bleeding complications:bleeding diathesis, thrombocytopenia (platelet count < 100 000/mm3), oral anticoagulant therapy (INR >1.6), uncontrolled hypertension (systolic blood pressure >200 mmHg), major bleeding, trauma or surgery within the last 30 days,
* acute renal failure,
* acute liver failure,
* pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-03; Primary Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
inhibition of platelet aggregation | at 30 days follow-up
  inhibition of platelet aggregation at the 30-day follow-up visit.
inhibition of platelet aggregation | at 1st hour after administration of the repeated loading dose of clopidogrel / placebo
  inhibition of platelet aggregation at 1st hour after administration of the repeated loading dose of clopidogrel / placebo
inhibition of platelet aggregation | at 2nd hour after administration of the repeated loading dose of clopidogrel / placebo
  inhibition of platelet aggregation at 2nd hour after administration of the repeated loading dose of clopidogrel / placebo
inhibition of platelet aggregation | at 6th hour after administration of the repeated loading dose of clopidogrel / placebo
  inhibition of platelet aggregation at 6th hour after administration of the repeated loading dose of clopidogrel / placebo
inhibition of platelet aggregation | at 24th hour after administration of the repeated loading dose of clopidogrel / placebo
  inhibition of platelet aggregation at 24th hour after administration of the repeated loading dose of clopidogrel / placebo

SECONDARY OUTCOMES:
Secondary outcome | 30 days
  frequency of bleeding complications within 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Roman Wojdyła, MD, Principal Investigator — Krakowskie Centrum Kardiologii Inwazyjnej, Elektroterapii i Angiologii Carint Scanmed Sp. z o.o
Locations (1):
- Krakowskie Centrum Kardiologii Inwazyjnej, Elektroterapii i Angiologii Carint Scanmed Sp. z o.o, Krakow, Poland